CLINICAL TRIAL: NCT01913990
Title: A Randomized, Phase IV Trial of Individualized Care Versus Standard Care, in the Prevention of Chemotherapy Induced Nausea and Vomiting in Breast Cancer Patients. The EPIC Study
Brief Title: Prevention of Chemotherapy Induced Nausea and Vomiting in Breast Cancer Patients.
Acronym: ER11-02
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011348-01H
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Emesis
Keywords: Nausea; Vomiting
MeSH Terms: conditions — Vomiting; Nausea | interventions — Dexamethasone; Ondansetron; Aprepitant; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Standard Anti-emetic regimen (Other): The standard anti-emetic arm:
  In this arm the treating medical oncologist will determine the choice of anti-emetic regimen that they perceive the patient would require and prescribe it. The treating physician will be blinded to result of the personalized composite emesis score. The physician may or may not choose to prescribe an NK-1 inhibitor as the study will not predetermine the type of anti-emetics used. In the event that the patient experienced chemo induced nausea and vomiting (CINV), modifications to the initial anti emetic regimen would be left to the treating physician.
  Interventions: Other: Arm A: Standard Anti-emetic regimen
- Arm B: Dexamethasone, Ondansetron, Aprepitant (Experimental): The emesis risk model arm:
  Prior to the start of intravenous chemotherapy an emesis risk score will be calculated for both acute and delayed emesis. The anti-emetic prophylaxis treatment will follow the emesis risk score. Whereby either an acute emesis score of ≥7 and/or a delayed emesis score of >16 will be considered high-risk. The anti-emetics will be prescribed reflecting this risk for pre-chemotherapy, 8 hrs post chemotherapy and day 2-3 post chemotherapy. Dexamethasone, Ondansetron and Aprepitant will be given in different combination and doses depending on what score the participant receives based on their responses to the diary. For subsequent cycle the anti-emetic score will be re-calculated prior to each cycle and the choice of anti-emetics adjusted if necessary.
  Interventions: Drug: Dexamethasone, Ondansetron, Aprepitant

INTERVENTIONS:
Drug: Dexamethasone, Ondansetron, Aprepitant — Arm B participants will be given doses of anti-emetics based on the emesis risk calculation. Doses will vary depending on the which level they fall into level 0, level 1, 2 or 3 based on the participant's diary.
  Other Names: Decadron; Zofran; Emend
  Arms: Arm B: Dexamethasone, Ondansetron, Aprepitant
Other: Arm A: Standard Anti-emetic regimen — Treating physician's discretion for type of anti-emetic to be prescribed.
  Arms: Arm A: Standard Anti-emetic regimen

SUMMARY:
For breast cancer patients receiving chemotherapy regimens, the use of a validated emesis (nausea and vomiting) risk calculator will provide superior anti-emetic (nausea and vomiting) control compared with "standard" anti-emetic regimen. The risk calculator has the potential to provide more individualized anti-emetic regimen by decreasing the use of toxic/costly anti-emetics in patients at low risk and possibly more importantly enhancing the appropriate anti-emetic regimen in patients at high risk.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed invasive breast cancer (stage I-III)

Scheduled to receive neoadjuvant or adjuvant intravenous anthracycline with cyclophosphamide-based chemotherapy;

Able to consent and fill study forms

Exclusion Criteria:

Received previous chemotherapy

Symptoms of nausea or vomiting at baseline (disease related)

On chronic anti-emetic therapy

On daily corticosteroids prior to initiation of chemotherapy

Allergic to steroids, 5HT3 or NK-1

Uncontrolled diabetes

Medical or psychiatric illness that would interfere with patients' ability to complete the diary

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of change in acute emesis (nausea and/or vomiting) in both study arms | Prior to each chemotherapy cycle every 3 weeks, at 24hrs post chemotherapy and at day 6 post chemotherapy for a total of 12 weeks
  The modified FLIE questionnaire is a patient-reported measure of the impact of chemotherapy induced emesis on daily life. It is a short, self administered instrument containing two domains-one for nausea (9 items) and one for vomiting (9 items). The modified FLIE questionnaire will be administered before the initiation of chemotherapy and on days 1 and 6, and prior to each cycle while on study. Responses to each question are scored on a 1- to 7-point scale as described in the FLIE Scoring Manual. For this study, "minimal or no impact of CINV on daily life" is defined as an average score of more than 6 on the 7-point scale. Additional data will be collected to assess physician anti-emetic prescribing habits as compared to published guidelines.

SECONDARY OUTCOMES:
Incidence of change in the delayed emesis (nausea and/or vomiting) in both study arms | Prior to each chemotherapy cycle every 3 weeks, at 24hrs post chemotherapy and at day 6 post chemotherapy for a total of 12 weeks
  The modified FLIE questionnaire is a patient-reported measure of the impact of chemotherapy induced emesis on daily life. It is a short, self administered instrument containing two domains-one for nausea (9 items) and one for vomiting (9 items). The modified FLIE questionnaire will be administered before the initiation of chemotherapy and on days 1 and 6, and prior to each cycle while on study. Responses to each question are scored on a 1- to 7-point scale as described in the FLIE Scoring Manual. For this study, "minimal or no impact of CINV on daily life" is defined as an average score of more than 6 on the 7-point scale. Additional data will be collected to assess physician anti-emetic prescribing habits as compared to published guidelines.

OTHER OUTCOMES:
Difference in breakthrough anti-emetic use in the emesis risk model group compared to the standard arm; i.e.: requirements for additional oral and parenteral anti-emetics during a single chemotherapy cycle | Prior to each chemotherapy cycle every 3 weeks, at 24hrs post chemotherapy and at day 6 post chemotherapy for a total of 12 weeks
  The modified FLIE questionnaire is a patient-reported measure of the impact of chemotherapy induced emesis on daily life. It is a short, self administered instrument containing two domains-one for nausea (9 items) and one for vomiting (9 items). The modified FLIE questionnaire will be administered before the initiation of chemotherapy and on days 1 and 6, and prior to each cycle while on study. Responses to each question are scored on a 1- to 7-point scale as described in the FLIE Scoring Manual. For this study, "minimal or no impact of CINV on daily life" is defined as an average score of more than 6 on the 7-point scale. Additional data will be collected to assess physician anti-emetic prescribing habits as compared to published guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, Dr., Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Clemons M, Bouganim N, Smith S, Mazzarello S, Vandermeer L, Segal R, Dent S, Gertler S, Song X, Wheatley-Price P, Dranitsaris G. Risk Model-Guided Antiemetic Prophylaxis vs Physician's Choice in Patients Receiving Chemotherapy for Early-Stage Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2016 Feb;2(2):225-31. doi: 10.1001/jamaoncol.2015.3730. PMID 26562292